CLINICAL TRIAL: NCT04873947
Title: Belun SpO2 Accuracy Comparison to Arterial Blood CO-Oximetry
Status: Completed | Type: Observational
Sponsor: Belun Technology Company Limited (Other)
Collaborators: Clinimark, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: PR2020-376
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- healthy adult volunteer: Subject is 18 to 50 years of age. Subject is a non-smoker or who has not smoked within 2 days prior to the study.
  Interventions: Device: Pulse Oximeter

INTERVENTIONS:
Device: Pulse Oximeter — The investigational device will be placed on the finger of the left or right hand per the instructions for use. Simultaneous data collection will be set up for the system under test and control oximeter.

SUMMARY:
This study was a comparative, single-center, non-randomized study conducted to evaluate the SpO2 accuracy per standards and guidelines identified above for SpO2 accuracy for pulse oximetry equipment over the range of 70-100% SaO2 under non-motion conditions. Arterial blood sampling measured by functional SaO2 CO-Oximetry, was used as the basis for comparison. Testing was conducted under normal office environment conditions.

DETAILED DESCRIPTION:
Pulse oximetry monitoring is considered a standard physiological measurement and is used by clinicians in everyday situations to estimate arterial oxygen saturation. A pulse oximeter is a device that measures the oxygen saturation of arterial blood non-invasively. In general, pulse oximeters use two wavelength absorption spectrophotometry to measure oxygen saturation based on the amount of reflected or scattered radiation. The wavelengths are selected to provide the best separation of absorbencies of oxy-hemoglobin (O2Hb) and deoxy-hemoglobin (HHb) states. The ratio of the two absorbencies is used to calculate the oxygen saturation (SpO2) value. Because an arterial sample of blood is not required to make the measurement, the pulse oximeter can provide non-invasive real time information. The clinical use of pulse oximeters has reduced the frequency and necessity of invasive arterial blood sampling, and has helped to improve patient safety by providing information to clinicians about patients' oxygenation status.

The purpose of this study was to evaluate the SpO2 accuracy performance of the Belun Ring Oximeter placed on the index fingers during non-motion conditions over the range of 70-100% SaO2 to arterial blood samples assessed by CO-Oximetry for an SpO2 validation.

The primary goal, was to show the SpO2 accuracy performance for the investigational device below. As a secondary goal, the pulse rate accuracy performance for the Belun ring was calculated.

It was expected that the Accuracy Root Mean Square (ARMS) performance would meet the required specification of ARMS 3.5% or lower in non-motion conditions for the range of 70 - 100% SaO2 thereby demonstrating an acceptable SpO2 accuracy performance specification. For the pulse rate accuracy, the desired goal was to have an accuracy performance of an ARMS of 3.

No risks or adverse device effects were expected. There were no contraindications for use in the proposed study / study population.

The study was conducted in accordance to the code of federal regulations for non-significant medical device studies and applicable ISO 14155 (2nd edition 2011-02-01), applicable sections of ISO 80601-2-61, second edition 2017-12, Corrected version 2018-02, and Pulse Oximeters - Premarket Notifications Submissions [510(k)s] Guidance For Industry and Food and Drug Administration Staff (issued: March 4, 2013).

ELIGIBILITY:
Inclusion Criteria:

* 10-15 Adults with a minimum of 3 males and a minimum of 3 females, with the balance made up of either
* Subject must have the ability to understand and provide written informed consent
* Subject is 18 to 50 years of age
* Subject must be willing and able to comply with study procedures and duration
* Subject is a non-smoker or who has not smoked within 2 days prior to the study

Exclusion Criteria:

* Subject is considered as being morbidly obese (defined as BMI >39.5)
* Compromised circulation, injury, or physical malformation of fingers, wrist, hands, ears or forehead/skull or other sensor sites which would limit the ability to test sites needed for the study. (Note: Certain malformations may still allow subjects to participate if the condition is noted and would not affect the particular sites utilized.)
* Female subjects that are actively trying to get pregnant or are pregnant (confirmed by positive urine pregnancy test unless the subject is known to be not of child-bearing potential).
* Smoker Subjects who have refrained will be screened for COHb levels >3% as assessed with a Masimo Radical 7 (Rainbow)
* Subjects with known respiratory conditions such as: (self-reported)

  * uncontrolled / severe asthma,
  * flu,
  * pneumonia / bronchitis,
  * shortness of breath / respiratory distress,
  * unresolved respiratory or lung surgery with continued indications of health issues,
  * emphysema, COPD, lung disease
* Subjects with known heart or cardiovascular conditions such as: (self-reported, except for blood pressure and ECG review)

  * hypertension: systolic >140mmHg, Diastolic >90mmHg on 3 consecutive readings (reviewed during health screen).
  * have had cardiovascular surgery
  * Chest pain (angina)
  * heart rhythms other than a normal sinus rhythm or with respiratory sinus arrhythmia (reviewed during health screen)
  * previous heart attack
  * blocked artery
  * unexplained shortness of breath
  * congestive heart failure (CHF)
  * history of stroke
  * transient ischemic attack
  * carotid artery disease
  * myocardial ischemia
  * myocardial infarction
  * cardiomyopathy
* Self-reported health conditions as identified in the Health Assessment Form (self-reported)

  * diabetes,
  * uncontrolled thyroid disease,
  * kidney disease / chronic renal impairment,
  * history of seizures (except childhood febrile seizures),
  * epilepsy,
  * history of unexplained syncope,
  * recent history of frequent migraine headaches,
  * recent symptomatic head injury (within the last 2 months)
  * cancer / chemotherapy
* Subjects with known clotting disorders (self-reported)

  * history of bleeding disorders or personal history of prolonged bleeding from injury
  * history of blood clots
  * hemophilia
  * current use of blood thinner: prescription or daily use of aspirin
* Subjects with severe contact allergies to standard adhesives, latex or other materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes or other medical sensors (self-reported)
* Subjects with severe allergies to iodine (only applicable if iodine is used)
* Subjects with severe allergies to lidocaine (or similar pharmacological agents, e.g. Novocain)
* Failure of the Perfusion Index Ulnar/Ulnar+Radial Ratio test (Ratio < 0.4)
* Unwillingness or inability to remove colored nail polish from test digits.
* Other known health condition, should be considered upon disclosure in health assessment form

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will include 10 to 15 healthy non-smoking (or has refrained from smoking for 2 days) competent adults, ages 18 to 50 years. The subject selection will be an equitable distribution of males and females of any race with varying skin tones including at least 2 darkly pigmented subjects or 15% of the subject pool, whichever is larger.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
Collect SpO2 data for accuracy statistical analysis by 10 subjects | 3 days
  Subjects were given medical grade mixtures of oxygen and nitrogen to induce stable plateaus across the range of 100% to 70%. The goal was to have an equal distribution of data by decade. The stable plateaus allowed data collection in the following SaO2 ranges 95-100, 90-95, 85-90, 80-85, 75-80, 70-75. In general, 4 to 8 discrete points were collected at each of the levels.
Accuracy data analysis | 3 days
  Data analysis follows ISO80601-2-61:2017, Annex EE and Pulse Oximeters - Premarket Notifications Submissions [510(k)s] Guidance For Industry and Food and Drug Administration Staff (issued: March 4, 2013).

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Cabrera, M.D., Principal Investigator — Clinimark, LLC
Locations (1):
- Clinimark, LLC, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No